CLINICAL TRIAL: NCT00290199
Title: A Randomized Controlled Trial of Foley Catheter for Labor Induction in Women With Term and Near Term Prelabor Rupture of Membranes (PROM)
Brief Title: Foley Catheter for Labor Induction in Women With Term and Near Term Membrane Rupture
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Gathering information from the PI records to provide this response.
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Alan Tita, Assoc Prof, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F051021005
Record Dates: First submitted 2006-02-09; First posted 2006-02-10 (Estimated); Results first posted 2012-10-31 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2017-04

CONDITIONS: Fetal Membranes, Premature Rupture; Labor, Induced/IS
Keywords: Fetal Membranes, Premature Rupture; Labor, Induced; Foley Catheter
MeSH Terms: conditions — Fetal Membranes, Premature Rupture

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transcervical Foley Catheter (Experimental)
  Interventions: Device: Transcervical Foley catheter
- No Foley (No Intervention)

INTERVENTIONS:
Device: Transcervical Foley catheter — Foley catheter placed through cervix for cervical ripening
  Arms: Transcervical Foley Catheter

SUMMARY:
In women undergoing labor induction for membrane rupture at or near term, we are investigating the addition of a foley catheter placed in the cervix to standard therapy (oxytocin administration) to decrease the time from the start of the induction to delivery.

DETAILED DESCRIPTION:
To compare the efficacy of a transcervical Foley catheter with concurrent oxytocin administration compared to oxytocin infusion alone for cervical ripening and labor induction in women with premature rupture of membranes (PROM) at > 34 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Preterm rupture of membranes (PROM) (Rupture of membranes = pooling/ferning/nitrazine +) Rupture of membranes (ROM) for ≥1 hour prior to starting induction
2. Cervix ≤ 2 centimeters (cm)
3. Gestational age ≥ 34 weeks by best obstetric estimate and clinical management decision is delivery
4. Singleton gestation
5. Cephalic
6. Vertex well applied to cervix

Exclusion Criteria:

1. Regular uterine contractions (contractions more frequent than every 5 minutes)
2. Two prior transverse uterine incisions/vertical uterine incision/ transmural myomectomy or any obstetric contraindication to labor
3. Evidence of chorioamnionitis (temperature of 100.4°F with uterine tenderness and maternal or fetal tachycardia or purulent discharge)
4. Lethal fetal anomalies
5. Intrauterine fetal demise (IUFD)
6. Previa
7. Suspected abruption/significant hemorrhage
8. Non-reassuring fetal heart rate (FHR) pattern
9. Non vertex fetal presentation

Ages: 12 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 169 (Actual)
Dates: Start 2005-12; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan T Tita, MD, Principal Investigator — University of Alabama at Birmingham
Locations (3):
- United States (3):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Christiana Care Health System, Newark, Delaware
  - Greenville Hospital System University Medical Center, Greenville, South Carolina

REFERENCES:
- [Background] Wolff K, Swahn ML, Westgren M. Balloon catheter for induction of labor in nulliparous women with prelabor rupture of the membranes at term. A preliminary report. Gynecol Obstet Invest. 1998;46(1):1-4. doi: 10.1159/000009986. PMID 9692332
- [Derived] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD001233. doi: 10.1002/14651858.CD001233.pub4. PMID 36996264

RESULTS

PARTICIPANT FLOW:
Groups:
- Transcervical Foley: Insertion of a foley catheter via the cervix prior to the initiation of induction with oxytocin
- No Foley: No insertion of a foley catheter via the cervix prior to the initiation of induction with oxytocin
Period: Overall Study
Arm/Group | Transcervical Foley | No Foley
Started | 87 | 82
Completed | 87 | 82
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Transcervical Foley | No Foley | Total
Number analyzed (Participants) | 87 | 82 | 169
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 87 | 82 | 169
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25 (5) | 25 (6) | 25 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87 | 82 | 169
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 87 | 82 | 169

OUTCOME MEASURES:

1. Primary Outcome: Hours From Placement of Foley or Initiation of Oxytocin to Delivery
Description: The outcome measure is the mean in hours of the time from induction to delivery (up to 24 hours)
Time Frame: Time from induction to delivery
Measure: Mean (Standard Deviation); unit: hours
Groups:
- Transcervical Foley: Insertion of a a transcervical foley catheter to induce labor
- No Foley: No transcervical foley catheter inserted to induce labor
Arm/Group | Transcervical Foley | No Foley
Number analyzed (Participants) | 79 | 73
hours | 10.8 (NA) — Due to PI no longer with institution, data not available | 12.1 (NA) — Due to PI no longer with institution, data not available.

2. Secondary Outcome: Rate of Delivery (Vaginal or Cesarean)by 24 Hours
Description: The percent of subjects having transcervical foley catheter and percent of subjects not having transcervical foley catheter delivering within 24 hours.
Time Frame: from start of induction to 24 hours post start of induction
Measure: Number; unit: percentage of deliveries
Arm/Group | Transcervical Foley | No Foley
Number analyzed (Participants) | 79 | 73
percentage of deliveries | 96 | 97

3. Secondary Outcome: Cesarean Rate
Description: The percent of subjects enrolled who had a cesarean at any time for any reason for delivery.
Time Frame: at delivery
Measure: Number; unit: percentage of subjects
Arm/Group | Transcervical Foley | No Foley
Number analyzed (Participants) | 79 | 73
percentage of subjects | 14 | 23

4. Secondary Outcome: Induction to Vaginal Delivery Interval
Description: Mean hours from time of induction to vaginal delivery interval.
Time Frame: time from induction to vaginal delivery, up to 24 hours
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Transcervical Foley | No Foley
Number analyzed (Participants) | 68 | 56
hours | 10.7 (NA) — Due to PI no longer with institution, data available. | 11.6 (NA) — Due to PI no longer with institution, data not available.

ADVERSE EVENTS:
Time Frame: From entry into study until delivery
Arm/Group | Transcervical Foley | No Foley
Serious Adverse Events (participants affected / at risk) | 0/87 | 0/82
Other Adverse Events (participants affected / at risk) | 0/87 | 0/82

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes